CLINICAL TRIAL: NCT02995187
Title: A Non-randomized, Open-label, Prospective, Single-center Study of Apatinib Mesylate Tablet as Third-line and Later Therapy in Patients With Small Cell Cancer（SCLC）
Brief Title: Study of Apatinib as Third-line and Later Therapy in Patients With Small Cell Lung Cancer (SCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yutao Liu, Associate Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-061
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Small Cell Lung Cancer
Keywords: Apatinib; Third-line and Later Therapy; Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib Mesylate tablet (Experimental): Patients received oral apatinib 500 mg in tablet once daily, a treatment cycle was defined as 28 days (4 weeks).
  Interventions: Drug: Apatinib Mesylate tablet

INTERVENTIONS:
Drug: Apatinib Mesylate tablet — Apatinib 500 mg in tablet once daily
  Other Names: Apatinib

SUMMARY:
This is a Single-center, Open-label, Single-arm,Non-randomized exploratory clinical trial evaluating the efficacy and safety of Apatinib for third-line and later treatment of patients with small cell lung cancer.

DETAILED DESCRIPTION:
Although fist-line therapy with Cisplatin and etoposide(EP)or Carboplatin and etoposide(CE)and second-line therapy with topotecan has been given, patients with extensive small cell lung cancer(ED-SCLC) still relapse and 2-year survival is less than 10%. There is no standard treatment recommendation for this group of patients who failed to second-line therapy and had good performance status. Apatinib has been approved as a second-line treatment for advanced gastric cancer. Several phase III clinical studies of non small cell lung cancer, liver cancer, colorectal cancer and other tumors also showed apatinib has less toxic side effects and better patient tolerance. However, the clinical application of apatinib in small cell lung cancer is still lack of evidence-based medicine. And this clinical trial is designed to prospectively investigate the efficacy and safety of apatinib in recurrent SCLC patients in our center.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 75 years;
2. Had a histologically or cytologically confirmed diagnosis of SCLC;
3. Had received at least 2 lines chemotherapy regimen and must include basis of the platinum regimen after which disease diagnosed;
4. Have not received VEGFR-TKI;
5. Had a life expectancy of at least 3 months;
6. Had an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2;
7. Had a disease status that was measurable or evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST, version1.1), larger than 10 mm in diameter by spiral CT scan;
8. Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥90g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, total bilirubin within 1.5×the upper limit of normal(ULN), and b) ALT and AST≤2.5×the ULN (If liver metastases, serum transaminase≤5×the ULN), serum creatine ≤ 1.25 x ULN, creatinine clearance rate > 45ml/min;
9. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug;
10. Signed and dated informed consent.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

1. Patients with non-small cell lung cancer;
2. Imaging (CT or MRI) results indicate that the existence of central tumors locally invading the large vessel could be detected, or apparent pulmonary cavity or necrotizing tumors;
3. Patients with clinical symptoms of brain metastases or meningeal metastasis;
4. Patients with poor-controlled arterial hypertension (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mm Hg) despite standard medical management;
5. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association (NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%;
6. Coagulant function abnormality (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT ULN > 1.5), with bleeding tendency or is treated with thrombolysis and anticoagulation;
7. Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g;
8. Patients who received major surgical operations or experienced severe traumatic injuries, bone fracture, or ulcers within 4 weeks before screening;
9. Patients who had obvious hemoptysis within 2 months before screening, or experienced daily hemoptysis with a volume more than half a tea spoon (2.5ml) or above; Patients who experienced bleeding symptoms of clinical significance , or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc;
10. Patients who manifested arterial/venous thrombus events, e.g.cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening;
11. Allergic to any ingredients of Apatinib;
12. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 3 years

SECONDARY OUTCOMES:
Overall survival | up to 3 years
Disease Control Rate | up to 3 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 3 years

OTHER OUTCOMES:
tumor phosphorylated VEGFR2 (p-VEGFR2) expressions | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yutao Liu, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Hu X, Jiang J, Yang L, Zhou S, Liu P, Li J, Wang Y, Hao X, Shi Y. A Prospective Study of Apatinib in Patients with Extensive-Stage Small Cell Lung Cancer After Failure of Two or More Lines of Chemotherapy. Oncologist. 2020 May;25(5):e833-e842. doi: 10.1634/theoncologist.2019-0391. Epub 2020 Apr 6. PMID 32250517